CLINICAL TRIAL: NCT04648722
Title: Higher Post-operative Levothyroxine Substitution Dose Needed in Right Compared to Left Lobe Hemithyroidectomy - a Retrospective Cohort Study
Brief Title: Higher Levothyroxine Requirements After Right-side Hemithyroidectomy
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Carola Deischinger, Principal investigator, Medical University of Vienna
Other Study IDs: Hemithyreoidectomy
Record Dates: First submitted 2020-11-22; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Hemithyroidectomy; Hypothyroidism
Keywords: Hemithyroidectomy; Levothyroxine; Postoperative levothyroxine requirements; Lobectomy; Thyroid
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Left-side hemithyroidectomy: Patients who received a hemithyroidectomy of the left thyroid lobe since 1994
  Interventions: Procedure: Hemithyroidectomy
- Right-side hemithyroidectomy: Patients who received a hemithyroidectomy of the right thyroid lobe since 1994
  Interventions: Procedure: Hemithyroidectomy

INTERVENTIONS:
Procedure: Hemithyroidectomy — We investigated patients who received a hemithyroidectomy at the Department of General Surgery, Division of Endocrine Surgery and a follow-up visit (3-12 months post-surgery) at the thyroid outpatient clinic of the Department of Endocrinology and Metabolism, Medical University of Vienna between 1994 and 2018.

SUMMARY:
459 adult patients who received a hemithyroidectomy at the Department of General Surgery, Division of Endocrine Surgery and a follow-up visit (3-12 months post-surgery) at the thyroid outpatient clinic of the Department of Endocrinology and Metabolism, Medical University of Vienna between 1994 and 2018 were identified and investigated in this retrospective study. The aim of this study was to investigate whether patients post right side hemithyroidectomy require a higher mean levothyroxine dosage than patients after left lobe hemithyroidectomy as the right thyroid lobe is bigger than the left lobe. Further, we aimed at developing a better post-surgery thyroid dosage prediction model.

DETAILED DESCRIPTION:
In most patients, the right lobe of the thyroid gland is larger than the left lobe. After a hemithyroidectomy, the remaining lobe grows by up to 30% to compensate for the loss. However, thyroxine replacement is still necessary for 22% to 60% of all patients. The aim of this study is to investigate whether a right-lobe hemithyroidectomy predisposes to a higher postoperative dose of levothyroxine.

Patients and Methods In a retrospective cohort study, 459 patients over the age of 18 years who underwent a hemithyroidectomy at the Department of General Surgery, Division of Endocrine Surgery and a follow-up (3-12 months post-surgery) visit at the thyroid outpatient clinic of the Department of Endocrinology and Metabolism between 1994 and 2018 were investigated. The study was approved by the local ethics committee and performed in accordance with the Declaration of Helsinki. The work has been reported in line with the STROCSS criteria. The patients were identified via data extraction from a university hospital-wide Research, Documentation and Analysis (RDA) database. In a second step, further information necessary for the analysis (ultrasound data on pre-surgery thyroid volume, pre-surgery TSH, side and date of hemithyroidectomy, surgery protocol, underlying thyroid disease, type and dosage of treatment, age, weight, height, thyrotropin (TSH), free T4 (fT4), free T3 (fT3)) were extracted from the internal electronic health record system. Patients who had either received radiation therapy had undergone previous thyroid surgery, surgery on the contralateral lobe, had pre-existing hypothyroidism, an autoimmune disease of the thyroid or were pregnant were excluded from the analysis. 33 patients were excluded due to additional surgery on the contralateral lobe resulting in a total of 426 patients. Pre-surgery ultrasound thyroid volume was calculated with the volumetric ellipsoid method (height × width × depth × correction factor 0.524).

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Males and females
* St.p. hemithyroidectomy

Exclusion Criteria:

* Radiation therapy
* Pregnancy
* Previous thyroid surgery (e.g. nodule removal surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who received a hemithyroidectomy at the Department of General Surgery, Division of Endocrine Surgery and a follow-up visit (3-12 months post-surgery) at the thyroid outpatient clinic of the Department of Endocrinology and Metabolism, Medical University of Vienna between 1994 and 2018 were identified and investigated in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Levothyroxine dosage | within 3 to 12 months post surgery
  dosage of levothyroxine needed post surgery, compared between left and right side hemithyroidectomy

SECONDARY OUTCOMES:
Hypothyroidism | within 3 to 12 months post surgery
  Incidence of hypothyroidism post surgery compared between left and right side hemithyroidectomy

CONTACTS AND LOCATIONS:
Overall Officials: Lana Kosi-Trebotic, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT04648722/Prot_SAP_000.pdf